CLINICAL TRIAL: NCT02495350
Title: The Correlation Between Prelabor Analgesic Plan and Actual Labor Analgesia With Satisfaction, Postpartum Depression, and Breast Feeding Success
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Dr. Sharon Orbach, Rabin Medical Center
Other Study IDs: 0666-14-RMC
Record Dates: First submitted 2015-06-17; First posted 2015-07-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Initially didn't want an epidural and didn't receive one.
- Initially didn't want an epidural and did receive one.
- Initially wanted an epidural and didn't received one
  Interventions: Other: Questionarie
- Initially wanted an epidural and did receive one.
  Interventions: Other: Questionarie

INTERVENTIONS:
Other: Questionarie — Parturients will be asked to fill out a labor satisfaction questionnaire detailing initial desire for epidural analgesia, final desire for epidural analgesia, adequacy of pain relief during labor and satisfaction with laborOn the third day postoperatively the parturients will be called and assessed for mood and signs of postpartum depression using Edinborough Postnatal Depression scale validated into Hebrew (10) , and we will assess whether or not they are breastfeeding.
  At 6 weeks we will follow-up to assess breastfeeding duration ,and postpartum depression using the Edinborough Postnatal Depression scale.
  Our comparison will include average pain scores, breast feeding success, and postpartum depression assessment.
  Groups: Initially wanted an epidural and did receive one.; Initially wanted an epidural and didn't received one

SUMMARY:
In this study the investigators would like to evaluate how prelabor analgesic plan and actual labor analgesia effects the labor satisfaction, breastfeeding success, and whether or not it reduces postpartum depression.

Although postpartum depression has been researched and reviewed, there is little information on how satisfaction during labor affects postpartum outcomes. The relationship between epidural analgesia is also complex, and there has yet to be found a valid correlation between the two parameters.

In addition although an attempt has been made to evaluate relationship between breastfeeding and epidural analgesia, results are unclear and further research is needed.

DETAILED DESCRIPTION:
This is a prospective, single center study, which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital.

All women undergoing vaginal delivery on the first day postpartum will be enrolled after filling out an informed consent.

They will be given out a labor satisfaction questionnaire detailing initial desire for epidural analgesia, final desire for epidural analgesia, adequacy of pain relief during labor and satisfaction with labor. (see appendix 1).

The investigators will evaluate breastfeeding success according to the latch scoring system in the first day postpartum which is routinely administered by nurses/ lactation consultants in the maternity ward.

According to their initial desire verses final analgesic choice they will be divided into four groups:

1. Women who initially didn't want and didn't receive one.
2. Initially didn't want and did receive one.
3. Initially wanted an epidural and didn't received one
4. Initially wanted an epidural and did receive one.

On the third day postoperatively the parturients will be called and assessed for mood and signs of postpartum depression using Edinborough Postnatal Depression scale validated into Hebrew (10) , and the investigators will assess whether or not they are breastfeeding.

At 6 weeks the investigators will follow-up to assess breastfeeding duration ,and postpartum depression using the Edinborough Postnatal Depression scale.

The investigators' comparison will include average pain scores, breast feeding success, and postpartum depression assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 undergoing vaginal delivery in Beilinson Hospital
* following obtaining written informed consents
* ability to comply with the study requirements will be included in the investigators' study

Exclusion Criteria:

* Women undergoing cesareans sections.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women above 18 undergoing vaginal delivery in Beilinson Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1954 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Assessment of postpartum depression using Edinborough Postnatal Depression scale | One year

SECONDARY OUTCOMES:
Assessment of breast feeding duration in women undergoing vaginal deliveries | one year
Increases in labor satisfaction defined as a vas (visual analog scale) satisfaction over 7 in women undergoing vaginal deliveries | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

REFERENCES:
- [Background] Hiltunen P, Raudaskoski T, Ebeling H, Moilanen I. Does pain relief during delivery decrease the risk of postnatal depression? Acta Obstet Gynecol Scand. 2004 Mar;83(3):257-61. doi: 10.1111/j.0001-6349.2004.0302.x. PMID 14995921
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Mauri PA, Contini NN, Giliberti S, Barretta F, Consonni D, Negri M, Di Benedetto I. Intrapartum epidural analgesia and onset of lactation: a prospective study in an Italian birth centre. Matern Child Health J. 2015 Mar;19(3):511-8. doi: 10.1007/s10995-014-1532-x. PMID 24894732
- [Background] Henderson JJ, Dickinson JE, Evans SF, McDonald SJ, Paech MJ. Impact of intrapartum epidural analgesia on breast-feeding duration. Aust N Z J Obstet Gynaecol. 2003 Oct;43(5):372-7. doi: 10.1046/j.0004-8666.2003.t01-1-00117.x. PMID 14717315
- [Background] Sheiner E, Shoham-Vardi I, Sheiner EK, Press F, Hackmon-Ram R, Mazor M, Katz M. A comparison between the effectiveness of epidural analgesia and parenteral pethidine during labor. Arch Gynecol Obstet. 2000 Feb;263(3):95-8. doi: 10.1007/s004040050003. PMID 10763834
- [Background] Dickinson JE, Paech MJ, McDonald SJ, Evans SF. Maternal satisfaction with childbirth and intrapartum analgesia in nulliparous labour. Aust N Z J Obstet Gynaecol. 2003 Dec;43(6):463-8. doi: 10.1046/j.0004-8666.2003.00152.x. PMID 14712952
- [Background] Kannan S, Jamison RN, Datta S. Maternal satisfaction and pain control in women electing natural childbirth. Reg Anesth Pain Med. 2001 Sep-Oct;26(5):468-72. doi: 10.1053/rapm.2001.24260. PMID 11561269
- [Background] Shapiro A, Fredman B, Zohar E, Olsfanger D, Jedeikin R. Delivery room analgesia: an analysis of maternal satisfaction. Int J Obstet Anesth. 1998 Oct;7(4):226-30. doi: 10.1016/s0959-289x(98)80043-5. PMID 15321184
- [Background] Glasser S, Barell V. [Depression scale for research in and identification of postpartum depression]. Harefuah. 1999 May 16;136(10):764-8, 844, 843. Hebrew. PMID 10955108
- [Background] Glasser S, Barell V, Shoham A, Ziv A, Boyko V, Lusky A, Hart S. Prospective study of postpartum depression in an Israeli cohort: prevalence, incidence and demographic risk factors. J Psychosom Obstet Gynaecol. 1998 Sep;19(3):155-64. doi: 10.3109/01674829809025693. PMID 9844846
- [Derived] Orbach-Zinger S, Landau R, Davis A, Oved O, Caspi L, Fireman S, Fein S, Ioscovich A, Bracco D, Hoshen M, Eidelman LA. The Effect of Labor Epidural Analgesia on Breastfeeding Outcomes: A Prospective Observational Cohort Study in a Mixed-Parity Cohort. Anesth Analg. 2019 Sep;129(3):784-791. doi: 10.1213/ANE.0000000000003442. PMID 31425221